CLINICAL TRIAL: NCT00409890
Title: The Effect of Hyoscine Butyl Bromide on the First Stage of Labor in Term Pregnancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital of the West Indies (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ECP 109,2004/2005
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Last update posted 2006-12-12 (Estimated); Status verified 2006-12

CONDITIONS: Labor Stage, First
Keywords: Buscopan; Hyoscine; Shortens; Labor; Stage

INTERVENTIONS:
Drug: Hyoscine Butyl Bromide

SUMMARY:
To determine whether hyoscine butyl bromide is effective in shortening the first stage of labor, with no increase in maternal or neonatal complications.

DETAILED DESCRIPTION:
Hyoscine butyl bromide has been used to shorten the duration of labor in several hospitals here in Jamaica, as it has elsewhere in the world. Thus, it represents a new addition to the armamentarium of active management. The mechanism by which it acts in the context of labor has not yet been elucidated, and the evidence for its efficacy was previously largely anecdotal. The specific objectives of this project are to assess whether hyoscine butyl bromide (in the form of Buscopan®) is effective in hastening cervical effacement and dilatation, thus shortening the duration of the first stage of labor. We also intend to determine whether the use of hyoscine butyl bromide in the first stage of labor has any associated increase in complications, such as an increase in blood loss or rate of Caesarean deliveries, or a decrease in neonatal APGAR scores.

The study was designed as a double blind, randomized, controlled, clinical trial comparing two groups of patients matched for age and parity. One group of patients received the 20 mg(1 ml)of hyoscine butyl bromide, while the other (control) group received 1 ml of normal saline (placebo).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Term pregnancy
* In spontaneous, established labour

Exclusion Criteria:

* Contraindication to vaginal delivery
* Any chronic medical or pregnancy induced illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-06; Study Completion 2005-10

PRIMARY OUTCOMES:
To assess whether hyoscine butyl bromide (in the form of Buscopan®) is effective in hastening cervical effacement and dilatation, thus shortening the duration of the first stage of labor.

SECONDARY OUTCOMES:
To determine whether the use of hyoscine butyl bromide in the first stage of labor has any associated increase in complications, such as an increase in blood loss or rate of Caesarean deliveries, or a decrease in neonatal APGAR scores.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Samuels, MD, Principal Investigator — University Hospital of the West Indies
Locations (1):
- University of the West Indies, Kingston, Kingston 7, Jamaica